CLINICAL TRIAL: NCT07220486
Title: Building Resilience in Skilled Nursing Care: A Behavioral Health Intervention for Residents & Care Partners
Brief Title: Behavioral Health Program for Short-Stay Nursing Facility Residents & Care Partners
Acronym: BRISK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Evan Plys, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P0001624; K23AG078410 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Nursing Home Resident; Skilled Nursing Facility; Depression; Feasibility Studies; Caregiver
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InSTILL (Experimental): Participants in this arm will participate in the Interventions for Stressful Transitions in Later Life (InSTILL), a behavioral health intervention tailored to the needs of short stay nursing facility residents and their primary care partner. InSTILL includes 8 sessions (2x per week for about 4 weeks) delivered in person or remotely. Both participants (e.g., resident and care partner) attend all sessions together, facilitated by a trained clinician.
  Interventions: Behavioral: Interventions for Stressful Transitions in Later Life
- Minimally Enhanced Usual Care (No Intervention): Participants in this group will receive a psychoeducational pamphlet with enhanced referrals for community support resources.

INTERVENTIONS:
Behavioral: Interventions for Stressful Transitions in Later Life — The Interventions for Stressful Transitions in Later Life (InSTILL) intervention is for skilled nursing facility residents and their care partners experiencing elevated levels of psychological distress. The intervention is designed to improve life management skills, emotion regulation skills, and dyadic coping skills with the goal of reducing depression symptoms among both dyad members (i.e., resident and care partner).
  Arms: InSTILL

SUMMARY:
The goal of this clinical trial is to test a behavioral health program (Interventions for Stressful Transitions in Later Life, InSTILL) for skilled nursing facility residents and their primary support person. The main questions it aims to answer is whether the program is program is feasible, satisfactory, and helpful. The researchers will compare the InSTILL program to minimally enhanced usual care. Participants will be randomly assigned to receive either the InSTILL program or minimally enhanced usual care. Participants will complete assessments at three timepoints (all) and a brief-exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient and care partner both aged ≥ 18 years
* Patient with care partner (known person providing regular health-related, socioemotional, or practical support) willing to participate
* Patient reporting depression symptoms on a screening tool (Patient Health Questionnaire)

Exclusion Criteria:

* Patient intended length of nursing facility stay < 7 days
* Patient evidencing more than mild impairment on a cognitive screen (Brief Interview for Mental Status)
* Patient's roommate in skilled nursing facility already enrolled in study/intervention
* Either patient or care partner reporting high risk of suicidality, based on a standardized safety assessment tool
* Either patient or care partner participating in newly initiated psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Credibility | peri-intervention
  3-item self-report measure of participant's belief regarding how helpful the intervention will be for them. Higher scores (min = 0, max = 30) scores indicate greater credibility.
Client Satisfaction Questionnaire | immediately after the intervention
  3-item self-report measure assessing patient satisfaction with the program. Higher total scores (min = 3, max = 12) indicate greater satisfaction.
Feasibility of Recruitment | baseline, pre-intervention
  Percentage of eligible approached dyads that are enrolled into the study.
Feasibility of Data Collection | 1 month follow-up
  Percentage of all participants with no measure fully missing at follow-up.
Treatment Adherence | immediately after the intervention
  Percentage of InSTILL participants completing 5/8 sessions
Clinician Fidelity | immediately after the intervention
  Percentage of InSTILL sessions delivered with 100% adherence on a study-specific Fidelity Checklist.
Adverse Events | 1 month follow-up
  Any adverse events related to participation in the study.
Treatment Acceptability Survey | immediately after the intervention
  Percentage of InSTILL participants scoring above the scale midpoint on all 9 Treatment Acceptability Survey items (developed for the current study).

SECONDARY OUTCOMES:
PHQ-9 | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  9-item self-report measure of depression symptoms. Higher scores (min=0, max=27) indicate greater depressive symptoms.
Selection, Optimization, and Compensation in Everyday Use | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  4-item self-report measure of the application of selection, optimization, and compensation strategies in daily life.
Committed Action Questionnaire | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  8-item self-report measure of pursuit of valued goals despite challenges and difficulties
Perceptions of Collaboration Questionnaire | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  12-item self-report measure of dyadic coping, including collaboration and interpersonal enjoyment.
General Anxiety Disorder-7 | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  7-item self-report measure of anxiety symptoms.
Euro QoL-5D 5L | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  6-item self-report measure of subjective health-related quality of life.
Relationship Assessment Scale | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  Single-item self-report measure of relationship satisfaction with study partner.
Preparedness for Future Care | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  5-item self-report measure of active preparation for future health care needs.
COREQ | immediately after the intervention
  4-item self-report of nursing facility satisfaction.
University of Washington Resilience Scale Short Form | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  4-item self-report of an individual's perceived resilience.
Zarit Burden Interview | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  4-item self-report screener of caregiver burden. Administered to care partners only.
Psychotropic medication use | baseline, pre-intervention; immediately after the intervention; 1 month follow-up
  Chart or self reported psychotropic medication use
Re-hospitalization | immediately after the intervention; 1 month follow-up
  Resident re-hospitalization during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Evan Plys, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No